CLINICAL TRIAL: NCT02537093
Title: A Pilot Study Examining Use of Asynchronous and Synchronous Telepsychiatry Consultation for Skilled Nursing Facility Residents
Brief Title: Pilot Study of Asynchronous and Synchronous Telepsychiatry for Skilled Nursing Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 741223
Record Dates: First submitted 2015-08-25; First posted 2015-09-01 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Dementia; Depression; Mood Disorder; Anxiety Disorder; Substance Use Disorder
MeSH Terms: conditions — Dementia; Depression; Mood Disorders; Anxiety Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synchronous telepsychiatry (STP) (Active Comparator): Control Arm/Synchronous telepsychiatry (STP): After baseline assessment, subjects will be assessed by a psychiatrist using live interactive videoconferencing every 6 months for a 1 year follow up (3 STP assessments: baseline plus 2 assessments). A report with treatment recommendations following American Psychiatric Association guidelines will be sent to the PCP who will be able to have adlib telephone or email consultations with the telepsychiatrist. The telepsychiatrist will have access to all previous clinical information about the patients.
  Interventions: Behavioral: Psychiatric Consultation
- Asynchronous telepsychiatry (ATP) (Experimental): Intervention Arm (ATP): All ATP assessments at 6 monthly intervals post baseline will be conducted by an ATP trained clinician. This interview will be video recorded.The ATP clinicians will then fill out a standardized medical template that will be reviewed by a psychiatrist who will provide a written assessment and psychiatric treatment plan. He will have access to any previous assessments and the PCP will also have continuing access to this psychiatrist by phone or email between the 3 consultations.
  Interventions: Behavioral: Psychiatric Consultation

INTERVENTIONS:
Behavioral: Psychiatric Consultation

SUMMARY:
Specific Aims: This study aims to assess the acceptability of asynchronous

telepsychiatry (ATP) and synchronous (STP) in rural Skilled Nursing Facility (SNF)

population, in a 12-month randomized controlled trial. ATP relies on video recording of a

psychiatric interview, where the video is later reviewed by a psychiatrist to make a

psychiatric diagnosis and treatment recommendation to the primary treatment team.

STP is real-time, face-to-face psychiatric assessment using video conferencing to come

up with a psychiatric recommendation. People residing in SNFs generally rely on primary

and consultant physicians to visit them and rarely have outpatient psychiatrist follow-up.

SNFs offer more services than what is available to primary care office, and include 24-

hours skilled nursing services, physical therapy, nutritional consultation, occupational

therapy, social services, wound care, and psychiatric consultation when available. SNF

residents are unable to live independently due to their multiple medical comorbidities

and are therefore more medically ill than patients who are typically seen in primary care

settings. The present study aims to demonstrate feasibility and to collect pilot data in

SNFs. This study is funded by the UC Davis Behavior Health Center of Excellence grant

via the California Mental Health Services Act (Prop 63). In a larger, future study, the investigators

intend to demonstrate that ATP will be no different than STP in clinical outcomes but will

be more accessible and cost effective.

DETAILED DESCRIPTION:
Specific Aims: This study aims to assess the acceptability of asynchronous

telepsychiatry (ATP) and synchronous (STP) in rural Skilled Nursing Facility

(SNF) population, in a 12-month randomized controlled trial. ATP relies on

video recording of a psychiatric interview, where the video is later reviewed by

a psychiatrist to make a psychiatric diagnosis and treatment recommendation

to the primary treatment team.

STP is real-time, face-to-face psychiatric assessment using video conferencing

to come up with a psychiatric recommendation. People residing in SNFs

generally rely on primary and consultant physicians to visit them and rarely

have outpatient psychiatrist follow-up. SNFs offer more services than what is

available to primary care office, and include 24-hours skilled nursing services,

physical therapy, nutritional consultation, occupational therapy, social services,

wound care, and psychiatric consultation when available. SNF residents are

unable to live independently due to their multiple medical comorbidities and are

therefore more medically ill than patients who are typically seen in primary care

settings. The present study aims to demonstrate feasibility and to collect pilot

data in SNFs. This study is funded by the University of California (UC Davis)

Behavior Health Center of Excellence grant via the California Mental Health

Services Act (Prop 63). In a larger, future study, we intend to demonstrate that

ATP will be no different than STP in clinical outcomes but will be more

accessible and cost effective.

Aim 1: To assess whether ATP and STP models improve clinical outcomes:

Hypotheses: Compared to STP, the ATP arm will: H1: show similar clinical

outcome trajectory, reflected in improvement from baseline, as measured by

Clinical Global Impression (CGI), Patient Health Questionaire-9 (PHQ-9), Brief

Interview for Mental Status (BIMS), and overall behavioral symptoms; H2: have

similar use of health care resources: psychiatric medications, additional interval

psychiatric visits, number of emergency room visits and hospitalizations

(medical, psychiatric, and overall); And H3: produce shorter waiting times for

psychiatric consultation.

Aim 2: To assess the acceptability of ATP and STP by examining satisfaction

surveys from SNF residents (who are able to complete the surveys).

Hypothesis:

Compared to STP, ATP participants will show: H1: Similar levels of satisfaction

as measured by: Telemedicine Satisfaction Survey as completed by

participants.

Aim 3: To conduct preliminary healthcare economics analysis and feasibility of

producing estimates of cost-effectiveness of ATP vs. STP in SNFs. Hypotheses:

ATP, compared to STP, will: H1: be more cost effective as measured by cost

savings from reduced need for face-to-face psychiatrist time and similar use of

other medical and psychiatric services.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18, with non-emergent psychiatric symptoms: depression, schizophrenia, bipolar disorder, Post-Traumatic Stress Disorder (PTSD), dementia-related behavioral problems, management of psychiatric medications, and other mental health problems that the Skilled Nursing Facility (SNF) Primary Care Provider (PCP) and team deems necessary to obtain psychiatric consultation.
* referred by SNF staff and PCP at participating site

Exclusion Criteria:

* Residents with imminent suicide and/or violence risks that require emergency psychiatric referrals or residents who cannot wait until the next ATP/STP evaluation
* Residents with other psychiatric emergencies will be referred to the local emergency department as is the current practice at both SNFs.
* less than 18 years
* immediate violent intentions or plans
* incarceration
* patient whose PCP recommends not participating.
* PCP not at participating site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression | 12 months
  Change in CGI will be measured from baseline to study endpoint of 12-month follow-up
Brief Interview for Mental Status (BIMS) | 12 months
  Change in BIMS will be measured from baseline to 12-month

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Norwood Pines Care Center, Sacramento, California
  - Cottonwood Post-Acute Rehabilitation Center, Woodland, California